CLINICAL TRIAL: NCT02034929
Title: A Randomized Controlled Study to Compare EndoCuff-assisted With Standard Colonoscopy for the Detection of Adenomas
Brief Title: EndoCuff-assisted Versus Standard Colonoscopy for Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Albert-Schweitzer-Klinik Northeim (Other)
Responsible Party: Principal Investigator, Tobias Meister, PD Dr. med., Helios Albert-Schweitzer-Klinik Northeim
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: HRS ID 003053
Record Dates: First submitted 2014-01-06; First posted 2014-01-14 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Polyp; Adenoma; Cancer
Keywords: colon cancer; adenoma; colon polyps
MeSH Terms: conditions — Polyps; Adenoma; Neoplasms; Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Endocuff-assisted colonoscopy (Active Comparator): Endocuff-assisted colonoscopy
  Interventions: Device: EndoCuff-assisted colonoscopy
- Standard colonoscopy (Active Comparator): Standard Colonoscopy
  Interventions: Device: Standard colonoscopy

INTERVENTIONS:
Device: EndoCuff-assisted colonoscopy — EC-assisted colonoscopy
  Arms: Endocuff-assisted colonoscopy
Device: Standard colonoscopy — Standard colonoscopy
  Arms: Standard colonoscopy

SUMMARY:
The EndoCuff is novel flexible cuff that can be attached to the distal tip of the colonoscope and helps to flatten large mucosal folds during withdrawal.

The study hypothesis is that the use of the Endocuff (EC) increases the adenoma detection rate during colonoscopy.

The study purpose is to compare EC-assisted colonoscopy with standard colonoscopy for polyp detection.

ELIGIBILITY:
Inclusion Criteria:

indication for colonoscopy (screening, surveillance, diagnostic) ager ≥ 18 years ability to give informed consent

Exclusion Criteria:

* pregnancy
* age<18 years
* known colonic strictures
* chronic inflammatory bowel disease
* active inflammation
* s/p colonic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | 25 minutes
  completion of colonoscopy is defined as the time point at which the colonoscope has been pulled out of the body.

SECONDARY OUTCOMES:
polyp detection rate | 1 Week
number of LGIN and HGIN adenomas detected | one week
  LGIN= low grade intraepithelial neoplasia HGIN= high grade intraepithelial neoplasia
polyp distribution | 25 minutes
procedure time | 25 Minutes
withdrawal time | 10 Minutes
  without intervention time due to polypectomy
ileum intubation rate | 10 minutes
total colonoscopy rate | 25 minutes
adverse events | 25 minutes
  perforation, cuff loss, lacerations, major bleedings, drop of sO2 during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, M.D., Principal Investigator — Helios Albert-Schweitzer-Hospital
Locations (4):
- Germany (4):
  - University Medical Center Göttingen, Göttingen
  - HELIOS St. Marienberg Hospital Helmstedt, Helmstedt
  - Helios Albert-Schweitzer-Hospital, Academic University Teaching Hospital, Northeim
  - HELIOS Medical Center Siegburg, Department of Gastroenterology, Siegburg

REFERENCES:
- [Derived] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133